CLINICAL TRIAL: NCT01482507
Title: Examination of the Effectiveness of Diffusion Weighted Magnetic Resonance Imaging for Identifying Poor Prognosis in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Optimus Clinical Research (Other)
Collaborators: Arthritis Australia, Abbott Australia (Unknown)
Responsible Party: Principal Investigator, Paul Bird, Principal Investigator, Optimus Clinical Research
Other Study IDs: IMM 10-0120 (DWI101)
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diffusion Weighted Imaging (DWI) MRI will assist in differentiating poor prognosis bone oedema more effectively than traditional T2 weighted MRI in patients with early Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
Assess DWI MRI in patients with early Rheumatoid Arthritis to determine whether the MRI method will assist in differentiating poor prognosis bone oedema more effectively than traditional T2 weighted MRI.

Aim 1: To compare DWI MRI with T2 weighted MRI for the discrimination of different types of bone oedema lesions in patients with early RA.

Aim 2: To examine the association between the presence of different types of bone oedema lesions detected on DWI MRI and T2 weighted MRI and the development of subsequent joint bone erosion as detected on i) MRI and ii) standard plain radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Rheumatoid Arthritis as defined by the ACR/Eular criteria
* Subject is able to understand and comply with study protocol
* Active disease as defined by DAS28> 3.0
* Disease duration less than 12 months
* If female, subject is either not of childbearing potential, or is of childbearing potential and is practicing an approved method of birth control throughout the study
* subject is judged to be in good health as determined by the PI based upon results of medical history, laboratory profile and physical examination.
* Prednisone dose 10mg or less, dose stable for 28 days prior to baseline

Exclusion Criteria:

* Inflammatory arthropathy other than Rheumatoid Arthritis
* Inactive disease as evidenced by DAS 28 CRP and / or ESR < 2.5
* Prednisone dose greater than 10mg within 28 days prior to baseline
* Intra-articular steroid within 28 days prior to baseline visit
* IV Methyl-prednisone within 28 days prior to baseline visit
* Any contra-indication to Magnetic Resonance Imaging
* Permanent Pacemaker
* Intracerebral aneurysm clip
* Claustrophobia to the extent that patient cannot manage MRI investigations
* Implanted metallic device
* Cochlear implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed Patients with active Rheumatoid Arthritis
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bird, Dr, Principal Investigator — Optimus Clinical Research
Locations (1):
- Optimus Clinical Research, Kogarah, New South Wales, Australia